CLINICAL TRIAL: NCT07366996
Title: Three-Dimensional Correction Methods for Idiopathic Scoliosis in Adolescent: Comparative Study
Brief Title: Three-Dimensional Correction Methods for Idiopathic Scoliosis in Adolescent
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Reda Rezk Nada, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005623
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Idiopathic Scoliosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schroth treatment (Experimental): Fifteen adolescents will participate in one-hour Schroth treatment sessions, conducted three times per week in center under therapist supervision on non-consecutive days.
  Interventions: Other: Schroth treatment
- Scientific Exercise Approach to Scoliosis (SEAS) (Experimental): The home program will consist of fifteen adolescents coming to the center once a month for Scientific Exercise Approach to Scoliosis (SEAS) treatment sessions, each lasting one hour. These sessions will be conducted three days per week, one hour, at home on non-consecutive days.
  Interventions: Other: Scientific Exercise Approach to Scoliosis (SEAS)

INTERVENTIONS:
Other: Schroth treatment — The exercise program targets three-dimensional spinal correction and includes Schroth breathing for rib cage expansion, pelvic tilts for pelvic alignment, side-shift exercises for lateral correction, rotational angular breathing for derotation, seated rotational stretches for lumbar flexibility, trunk elongation with resistance for postural strength, hanging stretches for spinal decompression, and arm-leg lifts to enhance core stability and coordination.
  Arms: Schroth treatment
Other: Scientific Exercise Approach to Scoliosis (SEAS) — The SEAS exercise program emphasizes active self-correction, core stability, and postural control during functional movements. Key exercises include pelvic tilts, seated forward bends, standing side bends, supine marching, bird-dog, heel slides, chest openers, and supine knee-to-chest stretches, all performed with self-correction to maintain neutral spinal alignment, improve muscular control, flexibility, and long-term postural stability.
  Arms: Scientific Exercise Approach to Scoliosis (SEAS)

SUMMARY:
This study aims to compare the effectiveness of "Schroth method" and "Scientific Exercise Approach to Scoliosis" for correcting idiopathic scoliosis in adolescents.

DETAILED DESCRIPTION:
The Schroth Method has gained prominence in the treatment of scoliosis due to its individualized approach, focusing on three-dimensional corrections through specific exercises tailored to each patient's spinal curvature. This method emphasizes rotational breathing and postural awareness, aiming to improve posture, reduce pain, and halt curve progression. Studies have shown that the Schroth Method can effectively improve spinal alignment, reduce curve severity, and enhance overall quality of life in patients with scoliosis. As a non-surgical intervention, it offers a valuable option for patients seeking to manage scoliosis conservatively. In contrast, the Scientific Exercise Approach to Scoliosis (SEAS) is another evidence-based method designed to treat scoliosis. SEAS focus on active self-correction, proprioceptive training, and functional exercises to stabilize and support the spine during daily activities. This approach is grounded in the principles of biomechanics and motor control, with an emphasis on developing the patient's ability to maintain correct posture independently. SEAS has been shown to be effective in reducing the risk of scoliosis progression and in some cases, it may reduce the need for bracing or surgery.

Comparing the Schroth Method and Scientific Exercise Approach to Scoliosis reveals significant insights into their respective benefits and limitations. While both approaches aim to address scoliosis through non-invasive means, they differ in their specific techniques and theoretical foundations. The Schroth Method's emphasis on breathing and postural correction contrasts with SEAS's focus on active self-correction and functional integration. Understanding these differences is crucial for clinicians to tailor treatment plans according to individual patient needs and preferences. This comparative study aims to provide deeper insights into the efficacy of these two approaches, potentially guiding more effective treatment strategies for adolescents with idiopathic scoliosis.

ELIGIBILITY:
Inclusion Criteria:

* Teenagers diagnosed with typical idiopathic scoliosis.
* Teenagers aged 13 to 18 years
* Both genders will be included.
* Participants with a Cobb angle ranging from 10° to 25°, as determined by radiographic analysis.
* Participants with Risser sign of 2 to 3, indicating incomplete skeletal maturity.
* Participants must be able to understand and follow instructions, ensuring effective participation in the treatment protocol.

Exclusion Criteria:

* Adolescents with significant visual or auditory impairments that could interfere with the ability to participate in or benefit from the rehabilitation programs.
* Adolescents with cognitive, mental, or psychological disorders that hinder understanding or following the instructions necessary for the treatment protocol.
* Adolescents who have previously undergone spinal surgery or any surgical interventions related to scoliosis or other spinal conditions.
* Adolescents with non-idiopathic scoliosis or scoliosis secondary to other underlying conditions (e.g., neuromuscular, congenital, or syndromic scoliosis).
* Adolescents with fixed spinal deformities that are not amenable to correction through non-surgical 3D approach.
* Adolescents with concurrent musculoskeletal conditions that could interfere with the treatment or assessment of scoliosis (e.g., significant hip or knee deformities).
* Adolescents currently participating in other clinical trials or receiving treatments that might confound the study results.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Cobb Angle | 12 weeks
  It will be assessed using standard standing posteroanterior spinal radiographs and will be measured before and after the intervention period. This outcome measure will be used to quantify the magnitude of the lateral spinal curvature and to evaluate changes in spinal alignment, allowing determination of the degree of curve correction or progression following the intervention.
Angle of Trunk Rotation (ATR) | 12 weeks
  It will be measured using a scoliometer during the Adam's forward bend test and will be assessed before and after the intervention period. This outcome measure will be used to evaluate the degree of rotational trunk deformity, reflecting the axial component of the three-dimensional spinal deformity in scoliosis.

SECONDARY OUTCOMES:
Risser Sign | 12 weeks
  It will be evaluated using pelvic radiographs and will serve as an indicator of skeletal maturity. This outcome measure will be used to estimate remaining growth potential and to assess the risk of scoliosis curve progression during the growth period.
Health-Related Quality of Life (HRQOL) | 12 weeks
  It will be assessed using validated Arabic versions of the Scoliosis Research Society-22 (SRS-22) questionnaire or the Pediatric Quality of Life Inventory (PedsQL). These instruments will be used to evaluate multiple domains affected by scoliosis, including pain, functional status, self-image, emotional well-being, and social functioning, providing a comprehensive measure of patients' perceived health and overall quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Olama, PhD, Study Chair — Professor, Cairo University; Maya Galal Abd El Wahab, PhD, Study Director — Ass. Professor, Cairo University
Locations (1):
- Faculty of Physical Therapy - Delta University for Science and Technology, Gamasa, Egypt